CLINICAL TRIAL: NCT07075328
Title: A Phase I/II Study of OJP-001 for Recurrent or Relapsed Adult T-cell Leukemia/Lymphoma Patients With Peripheral Blood Tumor.
Brief Title: A Phase I/II Study of OJP-001 in Patients With Adult T-cell Leukemia/Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Otsuka Medical Devices Co., Ltd. Japan (Industry)
Collaborators: JIMRO Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDT-21-001
Record Dates: First submitted 2025-06-27; First posted 2025-07-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-07

CONDITIONS: Adult T-Cell Leukemia/Lymphoma (ATLL)
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OJP-001 Group (Experimental): Patients will receive 5-ALA administered orally once. After administration of 5-ALA, patients will receive OJP-001 once.
  Interventions: Other: Drug:5-ALA, Device:Photodynamic system

INTERVENTIONS:
Other: Drug:5-ALA, Device:Photodynamic system — [Phase I part] Patients will receive 5-ALA administered orally once. After administration of 5-ALA, patients will receive Photodynamic system once.
  Dosage of 5-ALA: 10 mg/kg (1st cohort), 20 mg/kg (2nd cohort), 40 mg/kg (3rd cohort), 60 mg/kg (4th cohort) [Phase II part] Patients will receive 5-ALA and Photodynamic system once a week for 6 months.

SUMMARY:
This study aims to evaluate the tolerability of OJP-001, a therapeutic system combining photodynamic therapy (PDT) using OMD-001 and extracorporeal circulation therapy using OJE-001 and OJC-001, in patients with adult T-cell leukemia/lymphoma (ATL). The study will also investigate the recommended dose and pharmacokinetics of OMD-001, as well as the efficacy and safety of OJP-001.

DETAILED DESCRIPTION:
[Phase I part] Patients will receive 5-ALA administered orally once. After administration of 5-ALA, patients will receive OJP-001 once.

Dosage of 5-ALA: 10 mg/kg (1st cohort), 20 mg/kg (2nd cohort), 40 mg/kg (3rd cohort), 60 mg/kg (4th cohort)

[Phase II part] Patients will receive 5-ALA and OJP-001 once a week for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Hematocytologically or pathohistologically proven adult T-cell leukemia/lymphoma with positivity of anti-HTLV-1 antibody (Aggressive subtypes: acute, lymphoma type, or chronic type with unfavorable factor)
* Age: 20-85
* Meeting the any following criteria for screening

  * Relapsed or recurrent ATL have history of treatment with mogamulizumab
  * At least one regimen of chemotherapy in case of intolerance/contraindication for mogamulizumab
  * Relapsed or recurrent ATL judged inadequate of treatment with mogamulizumab by investigators
  * Relapsed or recurrent ATL after allogeneic hematopoietic stem cell transplantation
* Having peripheral blood lesion
* ECOG performance status: 0-2
* T-Bil: =< ULNx2, AST and ALT: =< ULNx2.5
* Expected more than 3 months of survival

Exclusion Criteria:

* Body Weight < 35kg
* Hemoglobin < 10g/dL
* Splenomegaly
* Subjects who received an following therapy

  * Chemotherapy or molecular-targeted agent for ATL : within 28 days prior to registration
  * Radiotherapy : within 28 days prior to registration
  * Any investigational drugs or medical devices (unapproved in Japan) : within 28 days prior to registration
  * Autologous stem cell transplantation : within 84 days prior to registration
  * Allogenic stem cell transplantation : within 100 days prior to registration
* Administrated 5-ALA drug except study drug within 7 days prior to registration
* Ate the foods containing 5-ALA or St. John's wort within 7 days prior to registration
* Synchronous or metachronous malignancy
* Uncontrolled severe complications
* Porphyria
* Uncontrolled cardiac arrhythmia or Chronic congestive heart failure (NYHA Class III or IV)
* Uncontrolled inter-current illness including: heart failure, kidney failure, liver failure, hypertension, diabetes mellitus
* Psychological disorder (mental illness, dementia, depression)
* HBs-Ag positive or HBc-Ab positive with HBV-DNA positive
* HCV-Ab positive
* HIV-Ab positive
* CNS involvement at screening
* QTcF > 470ms at screening
* Uncontrolled intercurrent infection
* Pregnant or nursing women
* During participated in other clinical trials
* Other inadequate conditions determined by investigators
* In phase II part: subjects who registrated in phase I part of this trial

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Phase I part: Dose limiting toxicity | Phase I part: 2 weeks
Phase II part: Response rate (best overall response) | Phase II part: 24 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Sapporo Hokuyu Hospital, Sapporo, Hokkaido
  - Imamura general hospital, Kagoshima, Kagoshima-ken
  - National Kyushu Cancer Center, Fukuoka
  - Nagasaki University Hospital, Nagasaki

IPD SHARING:
Plan to Share IPD: No